CLINICAL TRIAL: NCT07095478
Title: Phase II Single Arm, Open Label Study of Artesunate for the Treatment of Human Papilloma Virus Positive High Grade Cervical Intraepithelial Neoplasia (CIN2/3)
Brief Title: Safety and Efficacy of Oral Artesunate for Pre-cervical Cancer
Acronym: NeoART-CIN
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Metanoic Health Ltd. (Industry)
Collaborators: Clinical Research Malaysia (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-MHL-002; NMRR ID-24-01779-UWV (Other: National Medical Research Registration, Malaysia)
Record Dates: First submitted 2025-07-07; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: CIN 2/3
Keywords: CIN; HPV; drug repurposing; Artesunate; antimalarial
MeSH Terms: interventions — Artesunate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Artesunate (Experimental): 200mg oral tablets once daily for 14 days, with 7 days break for 3 cycles.
  Interventions: Drug: Artesunate

INTERVENTIONS:
Drug: Artesunate — Patients with HPV positive CIN2/3 will receive 3 cycles of oral artesunate 200mg OD prior to standard of care therapeutic LLETZ. Each 21 day treatment cycle will comprise oral artesunate 200mg OD for 14 days followed by a 7 day treatment break.

SUMMARY:
NeoART-CIN is a Phase II clinical study evaluating the safety and effectiveness of oral artesunate in patients with pre-cancerous cervical intra-epithelial neoplasia (CIN2/3), to investigate if a course of treatment with oral artesunate can reverse pre-cancerous changes in the cervix and prevent the development and progression of invasive cancer. Findings from this study will increase our understanding of the effects of artesunate on CIN2/3 and if confirmatory inform future clinical studies.

DETAILED DESCRIPTION:
Cervical cancer is the fourth most common form of cancer in women globally. It is a significant cause of morbidity and mortality, with over half a million new cases and over 300,000 deaths per year despite being preventable and curable if detected early and managed effectively. Low- and middle-income countries (LMICs) are disproportionately affected, with 80% of cases and 90% of cervical cancer-related deaths occurring in low-resource settings. There is an urgent need to develop affordable therapeutics to manage this global oncology burden. For many women, travel costs, time off work, and childcare responsibilities represent significant barriers to engaging with cervical cancer screening, treatment, and follow-up.

The World Health Organization (WHO) cervical cancer elimination strategy has set a target to eliminate cervical cancer as a public health problem (target incidence <4/100,000 population). To be on track to achieve this by the end of the century, draft targets include: 90% of girls vaccinated against HPV by the age of 15 years; 70% of all women aged 30 to 49 years receiving at least two high-precision screening tests 10 years apart; and 90% of screen-positive women, as well as 90% of women diagnosed with cervical cancer, receiving treatment by 2030. Countries are called to meet the 90-70-90 targets by 2030 in order to progress toward cervical cancer elimination. It is estimated that over 62 million deaths due to cervical cancer could be prevented in the next 100 years through implementation of this strategy alongside HPV vaccination.

While survival rates from colorectal, breast, prostate, cervical, and lung cancer are improving in high-income countries (HICs) due to a combination of early detection and more effective treatments, cancer death rates in LMICs are increasing. This is in part because many lifesaving cancer treatments remain unaffordable in LMICs, where cancer remains a neglected disease. Novel drug development takes an average of 10-15 years to go from bench to clinic at an average cost of USD 1 billion. Repurposing of established drugs for new indications can shorten this pathway substantially and reduce development costs.

In Malaysia, cervical cancer is the fourth leading cause of cancer-related morbidity and mortality among women, with an annual incidence of 1,700 cases reported in 2018. At present, only approximately 25% of women participate in regular cervical screening, and many patients present with advanced disease, with five-year overall survival around 52%. There is an urgent need for effective, safe, and affordable treatments to improve survival.

Artesunate belongs to the artemisinin family of sesquiterpene trioxane anti-malarial agents derived from Artemisia annua L. (Sweet wormwood), which has been used in traditional Chinese medicine for centuries to treat a variety of conditions including fever, inflammation, and haemorrhage. Artesunate is approved for the treatment of uncomplicated and multidrug-resistant malaria, is listed on the WHO Essential Medicines List, and is available at low cost (approximately USD 1 per daily dose).

Several comprehensive reviews have examined the anticancer effects of artemisinins. Pre-clinical studies in cell lines and animal models have demonstrated broad anticancer activity, including pro-apoptotic, anti-proliferative, anti-angiogenic, and anti-metastatic effects. A Phase I dose-escalation study of artesunate vaginal inserts in biopsy-confirmed cervical intraepithelial neoplasia (CIN) 2/3 in 28 participants demonstrated that treatment was safe and well tolerated, with histologic regression observed in 19 of 28 (67.9%) and HPV viral clearance in 9 of 19 (47.4%) participants. In participants who did not experience histological regression, no viral clearance was observed.

NeoART-CIN is a Phase II clinical study evaluating the safety and effectiveness of oral artesunate in participants with high-grade cervical intraepithelial neoplasia (CIN2/3), with the objective of determining whether a course of oral artesunate can reverse pre-cancerous cervical changes and prevent progression to invasive cancer. Findings from this study will increase scientific understanding of the effects of artesunate on CIN2/3 and may inform future clinical studies.

The primary research objective is to assess the feasibility, safety, and preliminary anti-proliferative activity of oral artesunate in HPV-positive high-grade CIN2/3.

A maximum of 28 participants will be enrolled to receive the study intervention. The primary endpoint is histological regression of CIN2/3, confirmed by colposcopy and biopsy at Day 90. The statistical design tests the null hypothesis that the response rate is 20%, versus the alternative that the response rate is 50%. The significance level is α=0.1, and the power is 90% when the true response rate is 50%. At a significance level of 0.05 and an equivalence margin of 0.15, a sample size of 24 participants is required to achieve 90% power, assuming a historical control response rate of 0.2 and an expected treatment response of 0.5. Accounting for a 20% loss to follow-up, the total sample size is inflated to approximately 28 participants.

Cervical cancer represents significant morbidity and mortality globally, particularly in LMICs. The current standard of care for women with high-grade CIN2/3 includes surgical or ablative treatments. Although these are generally safe, complications such as infection, bleeding, perforation, and cervical stenosis can occur. The most serious late complication is an increased risk of preterm birth and obstetric complications. Even after surgical resection with uninvolved margins, the risk of recurrence may range from 8% to 23%. For many women, barriers such as travel costs, time off work, and childcare continue to impede access to screening, treatment, and follow-up. There is an urgent need to develop safe, effective, and affordable therapeutics that can be delivered at the point of need. An oral treatment that is safe, effective, affordable, and capable of inducing regression of CIN2/3 and HPV clearance would represent a significant advance in the management of this condition.

Trial-specific risks and burdens include additional diagnostic, therapeutic, and monitoring procedures to assess safety, tolerability, and preliminary antiproliferative effects. Participants may not receive direct clinical benefit from participation, but their involvement will contribute to advancing scientific and clinical understanding of artesunate's potential role in treating CIN2/3.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or over
* Histologically proven HPV positive cervical CIN2/3
* WHO performance status 0-2
* Adequate full blood count:
* White Cell Count (WCC) >3.0 x 109 /l;
* Platelets >100 x 109/l;
* Haemoglobin (Hb) >80g/L
* Adequate renal function:
* Glomerular Filtration Rate >30ml/min
* Adequate hepatobiliary function:
* Total bilirubin < 3 x Upper limit normal
* Female participants of child bearing potential must have a negative pregnancy test < 72 hours prior to initiating study intervention and agree to avoid pregnancy using adequate, medically approved contraceptive precautions for up to 6 weeks after the last dose of study treatment intervention
* Patient able and willing to provide written, informed consent for the study

Exclusion Criteria:

* • Contraindication to the use of artesunate due to hypersensitivity

  * Pregnancy or lactation
  * Weight < 52 kg
  * History of previous CIN
  * Immunocompromised patients

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Histological regression of CIN2/3 on colposcopy and biopsy at Day 90 | From enrolment to end of trial at Day 90
  Histological regression will be defined as histologic regression to CIN1 or less.

SECONDARY OUTCOMES:
HPV DNA viral clearance at Day 90. | Measured at the end of the trial at Day 90
  Viral clearance will be defined as absence of HPV genotoype (s) detected at baseline.
Change in Vaginome Composition | At Day 1 , Day 64 of enrolment and at the end of the trial at Day 90
  Vaginal microbiota composition will be assessed using gene sequencing of vaginal swab samples collected at Day 1, Day 64, and Day 90. Changes in microbial diversity and relative abundance of dominant bacterial genera (e.g., Lactobacillus, Gardnerella) will be compared across time points. Microbial community structure will be analysed to evaluate shifts associated with the study intervention.
  Unit of Measure:
  Relative abundance (%), alpha diversity index, beta diversity distance metrics
Change in Gut Microbiome Composition Assessed | At Day 1 , Day 64 of enrolment and at the end of the trial at Day 90
  Gut microbiota composition will be assessed using gene sequencing of stool samples collected at Day 1, Day 64, and Day 90. Outcomes will include changes in relative abundance of dominant phyla (e.g., Firmicutes, Bacteroidetes), as well as measures of microbial diversity (alpha and beta diversity). Differences in community structure over time will be evaluated in relation to treatment exposure.
  Unit of Measure:
  Relative abundance (%), alpha diversity index, beta diversity distance metrics
Adverse events affecting patients as assessed by Common Terminology Criteria for Adverse Events (CTCAE) v5.0 | Assessment at Day 90 following study intervention
Patient-Reported Quality of Life (QoL) Assessed by Validated Questionnaires at Baseline | Assessment at Day 1 of study intervention (baseline)
  Quality of life will be assessed using validated, self-administered EQ- 5D-5L health questionnaire.
  Unit of Measure:
  Mean scores for each scale/domain of the EQ- 5D-5L questionnaires.
Patient-Reported Quality of Life (QoL) Assessed by Validated Questionnaires | Assessment at Day 7 of study intervention
  Quality of life will be assessed using validated, self-administered EQ- 5D-5L health questionnaire.
  Unit of Measure:
  Mean scores for each scale/domain of the EQ- 5D-5L questionnaires.
Patient-Reported Quality of Life (QoL) Assessed by Validated Questionnaires | Assessment at Day 14 of study intervention
  Quality of life will be assessed using validated, self-administered EQ- 5D-5L health questionnaire. Unit of Measure: Mean scores for each scale/domain of the EQ- 5D-5L questionnaires.
Patient-Reported Quality of Life (QoL) Assessed by Validated Questionnaires | Assessment at Day 22 of study intervention
  Quality of life will be assessed using validated, self-administered EQ- 5D-5L health questionnaire. Unit of Measure: Mean scores for each scale/domain of the EQ- 5D-5L questionnaires.
Patient-Reported Quality of Life (QoL) Assessed by Validated Questionnaires | Assessment at Day 43 of study intervention
  Quality of life will be assessed using validated, self-administered EQ- 5D-5L health questionnaire. Unit of Measure: Mean scores for each scale/domain of the EQ- 5D-5L questionnaires.
Patient-Reported Quality of Life (QoL) Assessed by Validated Questionnaires | Assessment at Day 64 of study intervention
  Quality of life will be assessed using validated, self-administered EQ- 5D-5L health questionnaire. Unit of Measure: Mean scores for each scale/domain of the EQ- 5D-5L questionnaires.
Patient-Reported Quality of Life (QoL) Assessed by Validated Questionnaires | Assessment at Day 90 of study intervention
  Quality of life will be assessed using validated, self-administered EQ- 5D-5L health questionnaire. Unit of Measure: Mean scores for each scale/domain of the EQ- 5D-5L questionnaires.
Change in Blood Biomarker Levels Associated with Cervical Intraepithelial Neoplasia (CIN 2/3) | Day 1, Day 14, Day 64, and Day 90
  Blood samples will be collected from participants with biopsy-confirmed CIN 2/3 at baseline (Day 1), Day 14, Day 64, and Day 90. Selected biomarkers relevant to HPV-related cervical dysplasia (e.g., pro-inflammatory cytokines such as IL-6, TNF-α, IFN-γ; and HPV-specific antibodies) will be quantified using validated immunoassays. The outcome will report changes in biomarker concentrations over time in relation to histological response.
  Unit of Measure:
  Concentration of biomarkers (e.g., pg/mL, IU/mL); fold-change from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Professor Sanjeev Krishna, FRCP, ScD, Study Chair — Centre of Diagnostics and Therapeutics; Dr Yolanda Augustin, Principal Investigator — Centre of Diagnostics and Therapeutics
Locations (5):
- Malaysia (5):
  - Pusat Perubatan Universiti Malaya, Kuala Lumpur, Kuala Lumpur
  - Institut Kanser Negara, Putrajaya, Kuala Lumpur
  - Hospital Umum Sarawak, Kuching, Sarawak
  - Hospital Ampang, Ampang, Selangor
  - Hospital Selayang, Batu Caves, Selangor

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF, CSR

REFERENCES:
- [Background] Liu Z, Zhang J, Li S, Jiang J. Artesunate Inhibits Renal Ischemia Reperfusion-Stimulated Lung Inflammation in Rats by Activating HO-1 Pathway. Inflammation. 2018 Feb;41(1):114-121. doi: 10.1007/s10753-017-0669-3. PMID 28921399
- [Background] Krishna S, Bustamante L, Haynes RK, Staines HM. Artemisinins: their growing importance in medicine. Trends Pharmacol Sci. 2008 Oct;29(10):520-7. doi: 10.1016/j.tips.2008.07.004. Epub 2008 Aug 25. PMID 18752857
- [Background] Kay J, Thadhani E, Samson L, Engelward B. Inflammation-induced DNA damage, mutations and cancer. DNA Repair (Amst). 2019 Nov;83:102673. doi: 10.1016/j.dnarep.2019.102673. Epub 2019 Jul 25. PMID 31387777
- [Background] Jansen FH, Adoubi I, J C KC, DE Cnodder T, Jansen N, Tschulakow A, Efferth T. First study of oral Artenimol-R in advanced cervical cancer: clinical benefit, tolerability and tumor markers. Anticancer Res. 2011 Dec;31(12):4417-22. PMID 22199309
- [Background] Ho WE, Peh HY, Chan TK, Wong WS. Artemisinins: pharmacological actions beyond anti-malarial. Pharmacol Ther. 2014 Apr;142(1):126-39. doi: 10.1016/j.pharmthera.2013.12.001. Epub 2013 Dec 6. PMID 24316259
- [Background] Heinonen A, Gissler M, Riska A, Paavonen J, Tapper AM, Jakobsson M. Loop electrosurgical excision procedure and the risk for preterm delivery. Obstet Gynecol. 2013 May;121(5):1063-1068. doi: 10.1097/AOG.0b013e31828caa31. PMID 23635744
- [Background] Hanahan D, Weinberg RA. Hallmarks of cancer: the next generation. Cell. 2011 Mar 4;144(5):646-74. doi: 10.1016/j.cell.2011.02.013. PMID 21376230
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Deeken JF, Wang H, Hartley M, Cheema AK, Smaglo B, Hwang JJ, He AR, Weiner LM, Marshall JL, Giaccone G, Liu S, Luecht J, Spiegel JY, Pishvaian MJ. A phase I study of intravenous artesunate in patients with advanced solid tumor malignancies. Cancer Chemother Pharmacol. 2018 Mar;81(3):587-596. doi: 10.1007/s00280-018-3533-8. Epub 2018 Feb 1. PMID 29392450
- [Background] Augustin Y, Staines HM, Krishna S. Artemisinins as a novel anti-cancer therapy: Targeting a global cancer pandemic through drug repurposing. Pharmacol Ther. 2020 Dec;216:107706. doi: 10.1016/j.pharmthera.2020.107706. Epub 2020 Oct 16. PMID 33075360

DOCUMENTS (1):
  • Study Protocol (2024-11-13): https://cdn.clinicaltrials.gov/large-docs/78/NCT07095478/Prot_000.pdf